CLINICAL TRIAL: NCT04359134
Title: Combined Evaluation of Pulmonary Fluids by Lung Ultrasounds and Transthoracic Electrical Bioimpedance in Preterm Infants With Respiratory Distress Syndrome
Brief Title: Combined Lung Ultrasounds and Transthoracic Electrical Bioimpedance in Preterm Infants With Respiratory Distress.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Niguarda Hospital (Other)
Responsible Party: Principal Investigator, Silvia Galletti, Assistant Researcher, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: Neo-POLM
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; Patent Ductus Arteriosus After Premature Birth; Perinatal Morbidity
Keywords: respiratory distress; patent ductus arteriosus; preterm infants; transthoracic electrical bioimpedance; lung ultrasounds
MeSH Terms: conditions — Dyspnea; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory distress syndrome (RDS) is among the most common complications of preterm birth, and typically becomes manifested soon after birth. A failure of the rapid reuptake of fetal lung fluids after birth, with subsequent liquid retention in the alveolar space, together with the deficit of surfactant proteins ensuing from lung immaturity represent the leading mechanisms for the development of RDS, which may require different levels of respiratory support.

An increasingly used method for the evaluation of the neonatal lung is pulmonary ultrasound, which allows assessing alveolar fluids and other pathological conditions in a non-invasive manner, and has been shown to predict the need for respiratory support and for surfactant administration in preterm infants with RDS. However, this method requires specific training, is operator-dependent and does not provide a trend able assessment over time.

Transthoracic electrical bioimpedance (TEB) allows continuous and non-invasive monitoring of static and dynamic thoracic fluids. It has been recently introduced in neonatal clinical practice to assess such hemodynamic parameters as cardiac output and also quantifies static thoracic fluids contents (TFC). This method provides continuous and non-operator dependent data on the pulmonary fluid status over time and does not require specific training.

The combination of lung ultrasound with TEB could open to new diagnostic and prognostic perspectives in preterm infants with RDS.

DETAILED DESCRIPTION:
Introduction Respiratory distress syndrome (RDS) is among the most common complications of preterm birth, and typically becomes manifested soon after birth. The rapid reuptake of fetal lung fluids plays an important role in transitional events at birth. Most of this fluid is reabsorbed through epithelial alveolar cells by an active sodium transporter. Mechanical events play a role in this exchange too. A failure of the rapid reuptake of fetal lung fluids after birth, with subsequent liquid retention in the alveolar space, together with the deficit of surfactant proteins ensuing from lung immaturity represent the leading mechanisms for the development of RDS, which may require different levels of respiratory support, ranging from mechanical ventilation to less invasive modalities (nasal cannulas or continuous positive airway pressure (CPAP)).

An increasingly used method for lung evaluation in the newborn is lung ultrasound, which allows to evaluate the alveolar fluid and to differentiate among several pathological conditions (transient tachypnea of the newborn, meconium aspiration, respiratory distress syndrome, pneumothorax, and pleural effusion) and, in the preterm population, has also been proved to predict of the need for respiratory support and for surfactant administration. Compared to traditional radiological assessments, this non-invasive technique does not imply the use of X-ray; however, it requires specific training, it is operator-dependent and does not allow a continuous and trend able evaluation over time, but only serial assessments.

Transthoracic electrical bioimpedance (TEB) allows continuous, non-invasive and real-time monitoring of static and dynamic thoracic fluids. It has been recently introduced in neonatal clinical practice to monitor such hemodynamic parameters as cardiac output, providing useful clinical information in hospitalized preterm infants, or neonates undergoing hemodynamic procedures. This technique allows quantifying static thoracic fluid contents (TFC) in a non-invasive and continuous manner. Compared to ultrasound, this method provides continuous and non-operator dependent data on the lung fluid status over time and does not require specific training for its use and interpretation.

Current literature reported a significant correlation between TFC values and respiratory distress, but, to date, it has not been investigated whether this parameter may predict RDS evolution, or if it is influenced by specific neonatal characteristics associated with pulmonary overflow, such as the presence of a patent ductus arteriosus (PDA), which is a common finding over the transitional period, defined as the first 72 hours of life.

Combining lung ultrasound to transthoracic electrical bioimpedance could open to new diagnostic and prognostic perspectives in preterm infants with RDS during the first days of life.

Objectives:

1. To evaluate the correlation between TFC, measured by transthoracic electrical bioimpedance (TEB), and a pulmonary ultrasound score, used for the evaluation of lung fluids in preterm infants with RDS in the Neonatal Intensive Care Unit.
2. To assess whether the combination of TFC with a pulmonary ultrasound score can be predictive of RDS evolution over the next 24 hours (need for surfactant, need for mechanical ventilation vs. suspension of ventilatory support).
3. Evaluation of pulmonary ultrasound score, TFC levels and left cardiac output in relation to the status of the ductus arteriosus (hemodynamically significant, restrictive or closed).

Methods:

Infants born at S. Orsola-Malpighi Hospital and Niguarda Hospital and admitted to the local Neonatal Intensive Care Units are consecutively enrolled in this observational prospective study if fulfilling the following eligibility criteria: gestational age ≤34 weeks' gestation, diagnosis of respiratory distress (defined by the need for respiratory support with nasal cannulas, nasal CPAP or mechanical ventilation), 0-24 hours of life, written informed consent obtained from parents/legal guardians of each infant.

The following conditions are considered as exclusion criteria: main congenital malformation, including congenital heart disease, meconium aspiration, pneumothorax, perinatal asphyxia/hypoxic-ischemic encephalopathy, concomitant use of experimental dugs.

Enrolled infants undergo serial lung and cardiac ultrasound evaluations at 0-24 (V1), at 24-48 (V2) and at 48-72 (V3)hours of life. A simultaneous evaluation of hemodynamic parameters and TFC by means of TEB is also performed.

Lung ultrasound findings are classified according to a validated pulmonary ultrasound score that takes into account six pulmonary fields (right upper anterior, right lower anterior, right lateral, left upper anterior, left lower anterior, left lateral). For each field a number is assigned:

* 0: only A lines or <3 B lines
* 1: ≥3 B lines
* 2: crowded and confluent B lines with or without consolidations
* 3: important consolidation If at 72 hours of life a hemodynamically relevant patent ductus arteriosus is still evident at cardiac ultrasound, the ultrasound and TEB monitoring are carried on until PDA closure.

Outcome: need for surfactant administration (and number of surfactant administrations), inhaled oxygen fraction, need for diuretic therapy, duration of ventilatory support with nasal canula/nasal CPAP/mechanical ventilation, duration of oxygen therapy, bronchopulmonary dysplasia at 36 weeks, duration of hospitalization and time for reach total enteral nutrition.

Statistic analysis: SPSS will be used for the statistical analysis. The diagnostic accuracy of TFC and of the ultrasound score for predicting the need for ventilatory support and for surfactant administration will be evaluated by area under ROC curve in order to find the optimal cut off value. The cardiac output values will be analyzed in relation to the state of the ductus arteriosus with Kruskal-Wallis test and included in a multivariate model in order to rule out the influence of confounding factors (for example the modality of ventilatory support). Significance level is set at p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* 0-24 hours of life,
* gestational age ≤34 weeks' gestation
* diagnosis of respiratory distress
* written informed consent obtained from parents/legal guardians of each infant.

Exclusion Criteria:

* major congenital malformations, including congenital heart disease
* meconium aspiration
* pneumothorax
* perinatal asphyxia/hypoxic-ischemic encephalopathy
* concomitant use of experimental drugs

Ages: 1 Day to 7 Days | Sex: All
Age Groups: Child
Study Population: Preterm infants ≤34 weeks' gestation with respiratory dystress
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between lung ultrasound score and RDS evolution | 0-24 hours of life
  Pearson correlation analysis between the score of lung ultrasound and RDS evolution over the next 24 hours (defined by the need for surfactant or a step-up in the type of respiratory support).
Correlation between lung ultrasound score and RDS evolution | 24-48 hours of life
  Pearson correlation analysis between the score of lung ultrasound and RDS evolution over the next 24 hours (defined by the need for surfactant or a step-up in the type of respiratory support).
Correlation between lung ultrasound score and RDS evolution | 48-72 hours of life
  Pearson correlation analysis between the score of lung ultrasound and RDS evolution over the next 24 hours (defined by the need for surfactant or a step-up in the type of respiratory support).
Correlation between TFC and RDS evolution | 0-24 hours of life
  Pearson correlation analysis between TFC values and RDS evolution over the next 24 hours (defined by the need for surfactant or a step-up in the type of respiratory support).
Correlation between TFC and RDS evolution | 24-48 hours of life
  Pearson correlation analysis between TFC values and RDS evolution over the next 24 hours (defined by the need for surfactant or a step-up in the type of respiratory support).
Correlation between TFC and RDS evolution | 48-72 hours of life
  Pearson correlation analysis between TFC values and RDS evolution over the next 24 hours (defined by the need for surfactant or a step-up in the type of respiratory support).
Correlation between TFC and lung ultrasound score | 0-24 hours of life
  Pearson correlation analysis between TFC values and lung ultrasound score
Correlation between TFC and lung ultrasound score | 24-48 hours of life
  Pearson correlation analysis between TFC values and lung ultrasound score
Correlation between TFC and lung ultrasound score | 48-72 hours of life
  Pearson correlation analysis between TFC values and lung ultrasound score

SECONDARY OUTCOMES:
Changes in TFC values and lung ultrasound score between time periods with patent and closed ductus arteriosus | 0-72 hours of life
  Changes in TFC and lung ultrasound scores between time periods with patent and closed ductus arteriosus

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Galletti, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi
Locations (2):
- Italy (2):
  - S. Orsola-Malpighi University Hospital, Bologna, Emilia-Romagna
  - Niguarda Hospital, Milan